CLINICAL TRIAL: NCT03832998
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Erenumab in Children (6 to < 12 Years) and Adolescents (12 to < 18 Years) With Chronic Migraine (OASIS PEDIATRIC [CM])
Brief Title: Efficacy and Safety of Erenumab in Pediatric Subjects With Chronic Migraine
Acronym: OASIS(CM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20160354; 2023-504928-26 (EudraCT Number); EMEA-001664-PIP02-15 (Other: EMEA)
Record Dates: First submitted 2019-01-29; First posted 2019-02-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Migraine; Headache; Prevention; Pediatric; Chronic Migraine
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1 (Experimental): Participants will be randomized to one of two doses determined by their body weight at Day 1. Participants who enrolled under the original protocol or protocol amendment 1 will be identified as group 1. Those enrolled under protocol amendment 2 will be identified as group 2.
  Interventions: Drug: Erenumab Dose 1; Drug: Erenumab Dose 2
- Dose Level 2 (Experimental): Participants will be randomized to one of two doses determined by their body-weight at Day 1. Participants who enrolled under the original protocol or protocol amendment 1 will be identified as group 1. Those enrolled under protocol amendment 2 will be identified as group 2.
  Interventions: Drug: Erenumab Dose 2; Drug: Erenumab Dose 3
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Erenumab Dose 1 — Participants in the low body-weight group at day 1 and who are randomized to Dose Level 1 will receive this dose.
  Other Names: AMG 334; Aimovig®
  Arms: Dose Level 1
Drug: Erenumab Dose 2 — Participants in the low body-weight group at day 1 who are randomized to Dose Level 2 and participants in the high body-weight group at day 1 who are randomized to Dose Level 1 will receive this dose.
  Other Names: AMG 334; Aimovig®
  Arms: Dose Level 1; Dose Level 2
Drug: Erenumab Dose 3 — Participants in the high body-weight group at day 1 who are randomized to Dose Level 2 will receive this dose.
  Other Names: AMG 334; Aimovig®
  Arms: Dose Level 2
Other: Placebo — Placebo matching dose for erenumab dose 1, 2 and 3.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of erenumab in migraine prevention in children (6 to <12 years) and adolescents (12 to <18 years) with chronic migraine. The study hypothesis is that in pediatric participants with chronic migraine, the combined erenumab dose group has a greater reduction from baseline to week 9 through week 12 (month 3) in monthly migraine days (MMDs) when compared with placebo in the double-blind treatment phase (DBTP).

DETAILED DESCRIPTION:
This study is a phase 3, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of erenumab in migraine prevention in children (6 to <12 years) and adolescents (12 to <18 years) with chronic migraine. The trial consists of four phases: screening (up to 3 weeks of initial screening and a 4-week prospective baseline phase); the DBTP (24 weeks for Group 1 subjects; 12-weeks for Group 2 subjects) in which participants receive placebo or erenumab dose 1, dose 2 or dose 3 (based on participant's body-weight) via subcutaneous injection once a month; the optional dose level blinded extension phase (40 weeks), in which all participants are assigned to receive dose 1, dose 2 or dose 3 of erenumab; and a 12 weeks safety follow-up phase (16 weeks after the last dose of investigational drug). The study intends to enrol 286 participants (256 adolescents and 30 children).

ELIGIBILITY:
Inclusion Criteria:

* Children (6 to less than 12 years of age) or adolescent (12 to less than 18 years of age) at the time of signing, if developmentally appropriate, the formal assent to participate to the study.
* Participant's parent or legal representative has provided written informed consent before initiation of any study-specific activities/procedures.
* History of migraine (with or without aura) for ≥ 12 months before screening according to the IHS Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2013) ICHD-3 specifications for pediatric migraine (participants aged less than 18 years), should be considered for the diagnosis of migraine.
* History of ≥ 15 headache days per month of which ≥ 8 headache days were assessed by the participant as migraine days per month in each of the 3 months prior to screening.
* Migraine frequency: greater than or equal to 8 migraine days based on the eDiary data during the last 28 days of the baseline phase if more than 28 days in duration.
* Headache frequency of greater than or equal to 15 headache days based on the eDiary data during the last 28 days of the baseline phase if more than 28 days in duration.
* Demonstrated at least 80% compliance with the eDiary based on the last 28 days of the baseline period, if more than 28 days in duration (eg, completing eDiary items for at least 23 out of the last 28 days of the baseline phase).

Key Exclusion Criteria:

* History of cluster headache or hemiplegic migraine headache.
* Chronic migraine with continuous pain, in which the participant does not have any pain free periods (of any duration) during the 1 month prior to screening.
* No therapeutic response with greater than 3 medication categories for prophylactic treatment of migraine after an adequate therapeutic trial. No therapeutic response is defined as no reduction in headache frequency, duration, or severity after administration of the medication for at least 6 weeks at the generally-accepted therapeutic dose(s) based on the investigator's assessment.
* History of suicidal behavior or the participant is at risk of self-harm or harm to others.
* History of major psychiatric disorder. Participants with anxiety disorder and/or mild major depressive disorder (Patient Health Questionnaire Modified for Adolescents [PHQ-A] score 9 for adolescents or based on medical judgement of the investigator for children) are permitted in the study if they are considered by the investigator to be stable and are taking no more than 1 medication for each disorder. Participants must have been on a stable dose within the 3 months before the start of the baseline phase.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in MMDs | Baseline through week 12 of DBTP
  To evaluate the effect of erenumab compared with placebo on the change in MMDs from baseline to week 9 through week 12 (month 3) of DBTP.

SECONDARY OUTCOMES:
Change in monthly headache days from baseline | Baseline through week 12 of the DBTP
  To evaluate the effect of erenumab compared with placebo on the change from baseline in monthly headache days to week 9 through week 12 (month 3) of DBTP.
Proportion of participants with at least 50% reduction in MMDs from baseline | Baseline through week 12 of the DBTP
  To evaluate the effect of erenumab compared with placebo on the proportion of participants with at least 50% reduction in MMDs from baseline to week 9 through week 12 (month 3) of the DBTP.
Change in MMDs from baseline to the average of the first 3 months | Baseline through week 12 of the DBTP
  To evaluate the effect of erenumab compared with placebo on the change in MMDs from baseline to the average of the first 3 months (week 1 through week 12) of the DBTP.
Change in monthly average severity of migraine attacks from baseline (measured with a visual analogue scale) | Baseline through week 12 of the double blind treatment phase
  To evaluate the effect of erenumab compared with placebo on the change from baseline in monthly average severity of migraine attacks to week 9 through week 12 (month 3) of the DBTP. This will be measured in an electronic diary (eDiary) with a visual analogue scale.
Change from baseline in migraine-related disability and productivity as assessed by the Pediatric Migraine Disability Assessment (PedMIDAS) | Baseline through week 12 of the DBTP
  To evaluate the effect of erenumab compared with placebo on the change from baseline in migraine-related disability and productivity as measured by the modified PedMIDAS to week 9 through week 12 (month 3) of the DBTP.
Number of participants experiencing Treatment-emergent Adverse Events (TEAE) | Up to Week 83
  TEAEs are any event that occurred after the participant received study treatment. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occurred after study treatment administration were recorded as TEAEs. A serious TEAE is any untoward medical occurrence in a clinical study participant after first dose irrespective of a causal relationship with the study treatment(s) that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
Number of participants expressing C Terminal Telopeptide of Type 1 Collagen (CTX) Markers | Up to week 83
Number of participants expressing Procollagen Type 1 N Propeptide (P1NP) Markers | Up to week 83
Number of participants expressing Anti-erenumab antibodies | Up to week 83
Change in growth and development rate as assessed by physical measuraments based on age-adjusted Z-scores for height and weight | Up to week 83
Number of participants experiencing treatment-emergent suicidal ideation and behavior as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS). | Up to week 83
Group 1 only: Number of participants experiencing injection site pain as assessed by Face Pain Scale-revised (FPS-R) | Day 1 and week 20
Group 2 only: Number of participants experiencing injection site pain as assessed by FPS-R | Day 1 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (101):
- United States (38):
  - Paradigm Clinical Research Center Inc, San Diego, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Childrens National Health System, Washington D.C., District of Columbia
  - TrueBlue Clinical Research, Brandon, Florida
  - Northwest Florida Clinical Research Group Limited Liability Company, Gulf Breeze, Florida
  - Nicklaus Childrens Hospital, Miami, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Rare Disease Research Center Pediatrics, Atlanta, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Chicago Headache Center and Research Institute, Chicago, Illinois
  - Josephson Wallack Munshower Neurology, Indianapolis, Indiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - New England Regional Headache Center Inc, Worcester, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute Inc, Plymouth, Minnesota
  - Childrens Mercy Hospital and Clinics, Kansas City, Missouri
  - Mercy Research, St Louis, Missouri
  - Meridian Clinical Research LLC, Hastings, Nebraska
  - Dent Neurosciences Research Center, Amherst, New York
  - Modern Migraine MD, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Inc, Pittsburgh, Pennsylvania
  - Palmetto Gastroenterology Clinical Research, LLC, Summerville, South Carolina
  - Child Neurology Consultants of Austin, Austin, Texas
  - Helios Clinical Research Inc, Burleson, Texas
  - Stryde Consulting LLC, Frisco, Texas
  - Childrens Specialty Group, Norfolk, Virginia
  - Vaught Neurological Services, Crab Orchard, West Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels
  - Algemeen Ziekenhuis Sint-Maarten, Mechelen
  - Docteur Simona Sava, Saint-Nicolas
- Canada (4):
  - Stollery Childrens Hospital, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital For Sick Children, Toronto, Ontario
- Colombia (3):
  - Fundacion Centro de Investigacion Clinica, Medellín, Antioquia
  - Cafam, Bogota, Cundinamarca
  - Fundacion Cardiovascular de Colombia, Bucaramanga, Santander Department
- Terveystalo Pulssi, Turku, Finland
- Germany (4):
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Universitaetsklinikum Essen, Essen
  - Schmerzklinik Kiel, Kiel
  - Arzneimittelforschung Leipzig GmbH, Leipzig
- Hungary (6):
  - Dr Kenessey Albert Korhaz - Rendelointezet, Balassagyarmat
  - Dr Altmann Anna egyeni vallalkozo, Budapest
  - High Tech Medical Kft, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
- Italy (4):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda di Rilievo Nazionale e Alta Specializzazione Civico Di Cristina Benfratelli, Palermo
  - Fondazione Istituto Neurologico Nazionale C Mondino IRCCS, Pavia
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
- Japan (16):
  - Josai Kids Clinic, Nagoya, Aichi-ken
  - Medical Corporation Seikokai Takanoko Hospital, Matsuyama, Ehime
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - Kitami Clinic, Sapporo, Hokkaido
  - Konan Medical Center, Kobe, Hyōgo
  - Kumamoto City Hospital, Kumamoto, Kumamoto
  - Tatsuoka Neurology Clinic, Kyoto, Kyoto
  - Japanese Red Cross Kyoto Daiichi Hospital, Kyoto, Kyoto
  - Sendai Headache and Neurology Clinic, Sendai, Miyagi
  - Tominaga Hospital, Osaka, Osaka
  - Saitama Neuropsychiatric Institute, Saitama-shi, Saitama
  - Tokyo Headache Clinic, Shibuya-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Nagamitsu Clinic, Hofu-shi, Yamaguchi
  - Nagaseki Headache Clinic, Kai-shi, Yamanashi
- Poland (9):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Centrum Medyczne Luxmed Spzoo, Lublin
  - Centrum Medyczne Hope Clinic Sebastian Szklener, Lublin
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Clinical Research Center Spzoo Medic-R Spolka Komandytowa, Poznan
  - Dr Sekowska Leczenie Bolu, Warsaw
  - Next Stage Spzoo, Warsaw
  - Migre Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw
- Puerto Rico Health and Wellness Institute, Dorado, Puerto Rico
- Russia (4):
  - FSBI Russian Children Clinical Hospital of the MoH RF, Moscow
  - LLC clinic Chaika, Moscow
  - LLC Sibneyromed, Novosibirsk
  - LLC Medical Technologies, Saint Petersburg
- United Kingdom (8):
  - Noahs Ark Childrens Hospital for Wales, Cardiff
  - Royal Hospital for Children, Glasgow
  - 4 Medical Clinical Solutions London, Ilford
  - Alder Hey Childrens Hospital, Liverpool
  - Evelina Childrens Hospital, London
  - Great Ormond Street Hospital for Children, London
  - 4 Medical Clinical Solutions Manchester, Manchester
  - Oxford Childrens Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com